CLINICAL TRIAL: NCT00364364
Title: Pharmacokinetics, Biodistribution and Targeting of 111 In- Labeled Humanized PAM4IgG in Pre-Surgical Pancreatic Cancer Patients.An Examination of Protein Dose
Brief Title: Safety Study to Determine the Appropriate Dose of Antibody Against Tumor Cells to Best Target Patients With Pancreatic Cancer.
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0473; CA098488; 05-02-07-05 (Other: JHM IRB); C-062B-03 (Registry Identifier: NCI)
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2008-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

INTERVENTIONS:
Drug: Radiolabeled humanized PAM4 IgG

SUMMARY:
This no treatment research study is being done to find a safe and an appropriate dose of antibody (protein) against tumor cells to best target the cancer in people with pancreatic cancer. To do this, this no-treatment research study will compare two doses of an antibody called hPAM4 IgG when combined with a radioactive element, Indium-111.

DETAILED DESCRIPTION:
This is an open-label, single-center, non-randomized, single-arm, pilot imaging study to determine the pharmacokinetics, biodistribution, and tumor targeting of an indium-111 (111In)-labeled, humanized anti-MUC1 antibody, designated hPAM4 IgG1 in patients with known pancreatic cancer. The primary objective of this trial is to examine how changing the protein dose will affect these parameters with the intent to determine if a single protein dose can be selected to optimize tumor targeting. It is expected that these data will aid in the selection of an appropriate protein dose to be used in a Phase I therapy trial with yttrium-90 (90Y)-labeled hPAM4 IgG. The secondary objective is to monitor safety.

Pharmacokinetics, biodistribution, tumor targeting, and dosimetry (modeling for 90Y) will be assessed against clinical parameters, such as pre-study PAM4-reactive MUC-1 antigen in the serum, tumor size, location, histopathology, immunohistology, and if possible, antigen content by extraction of tumor sample.

ELIGIBILITY:
Inclusion Criteria:-

* All patients must either have a histologic or cytological diagnosis of pancreatic cancer or a high clinical suspicion of pancreatic cancer.
* Patients must be 21 years of age.
* Patients must have measurable disease by CT scan.
* Patients must be at least 4 weeks beyond any major surgery.
* Patients must be at least 4 weeks beyond any chemotherapy or radiation therapy and must have recovered from treatment-induced toxicity.
* Patients must have a performance status of 70% or greater on the Karnofsky Scale and a minimal life expectancy of 3 months.
* Patients must not have severe anorexia, nausea or vomiting, and no signs of intestinal obstruction.
* Patients must have a serum creatinine that is < 1.5 x the Institutional Upper Limit of Normal (IULN).
* AST/ALT < 2 times the IULN; serum bilirubin < 3 x IULN.
* WBC 3000/mm3, a granulocyte count 1500/mm3, and a platelet count 100,000/mm3.
* Patients must sign an informed consent, and be mentally responsible. There will be no discrimination based on race, creed, or ethnic background.
* Patients must be able to return to an approved study site for the scheduled follow-up procedures.

Exclusion Criteria:

A.Subjects with a significant concurrent medical complication that in the judgment of the Principal Investigator could affect the patient's ability to tolerate or complete this study. These include, but are not restricted to

1. Known history of active coronary artery disease, unstable angina, myocardial infarction, or congestive heart failure present within 6 months or cardiac arrhythmia requiring anti-arrhythmia therapy.
2. Known history of active COPD, or other moderate-to-severe respiratory illness present within 6 months.

B. Subjects who have signs of intestinal obstruction.

C. Subjects who are pregnant are excluded. D. Subjects who have a measurable antibody response to hPAM4 in their pre-study sample or who are proven allergic upon testing with the agent.

E. Patients who are known to have HIV.

F. Patients who have a known history of Hepatitis B or C or any other serious liver abnormality will be excluded from enrollment.

G. Prisoners or other institutionalized persons.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Examine the pharmacokinetics and tumor targeting of 111In-DOTA-hPAM4 anti-MUC-1 IgG given intravenously to patients with known or a suspicion of primary or recurrent pancreatic cancer.
An examination of how the pharmacokinetics and tumor targeting are affected by the amount of hPAM4 IgG administered.
Targeting with 111In-hPAM4 will be compared to other radiological (e.g., CT) and nuclear (FDG-PET; optional)findings.
For patients who undergo surgery after the 111In-hPAM4 study, targeting will be correlated against surgical findings.

SECONDARY OUTCOMES:
Correlate tumor targeting, when feasible, with the following:Immunohistology using the hPAM4 antibody
Histology,Serum antigen content
Determine normal organ and, whenever possible, tumor dosimetry for 90Y-hPAM4 IgG based on the distribution and tumor targeting of 111In-hPAM4-IgG.
Monitor the development of antibody formation to the hPAM4, when feasible.
Targeting with 111In-hPAM4 will be compared to other radiological (e.g., CT) and nuclear (FDG-PET; optional)findings.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wahl, MD, Principal Investigator — Johns Hopkins Institution
Locations (1):
- Johns Hopkins Institution, Dept of Radiology and Radiological Science, Baltimore, Maryland, United States